CLINICAL TRIAL: NCT03337659
Title: Child Developmental Health, Maternal Psychosocial Distress, and Health System Costs At 18 Months Corrected Age: Effectiveness of a Cluster Randomized Controlled Trial of Family Integrated Care in Level II NICUs
Brief Title: A Cluster Randomized Controlled Trial of FICare At 18 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other); University of Alberta (Other); Alberta Health services (Other)
Responsible Party: Principal Investigator, Karen Benzies, Professor; Associate Dean, Research, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CIP-150740
Record Dates: First submitted 2017-10-23; First posted 2017-11-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2020-11

CONDITIONS: Premature Birth
Keywords: Family-integrated care; neonatal intensive care unit; premature; infant development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FICare Intervention Group (Experimental): Study participants received Family Integrated Care (intervention) while their infant(s) was/were admitted to a Level II NICU.
  Interventions: Other: Family Integrated Care
- FICare Control Group (No Intervention): Study participants received standard care while their infant(s) was/were admitted to a Level II NICU.

INTERVENTIONS:
Other: Family Integrated Care — FICare is a dynamic psycho-educational intervention. The goal of FICare is a change in culture and practice that permits, encourages and supports parents in their parenting role while their infant is receiving health care in a Level II NICU. Underpinned by adult learning and change theories, FICare empowers parents to build their knowledge, skill and confidence so that the family is well-prepared to care for their infant long before discharge.
  Other Names: FICare
  Arms: FICare Intervention Group

SUMMARY:
In Alberta, one in every twelve babies is born preterm. Compared with their full term counterparts, preterm infants who survive are at higher risk for respiratory problems, jaundice, infections, feeding problems, behavioural problems, and neuro-developmental disabilities, including cognitive delays, and visual and hearing impairments. As a result, parents must leave their preterm babies in the hospital to fully develop enough to care for them at home. When it is time for discharge, parents are often unprepared to look after their baby because they may have limited involvement in the care of their baby in hospital. In addition to the distress and costs to parents of having a baby in hospital, health system costs are also increased the longer a baby is in hospital. The aim of this novel health services study is to assess the longer-term outcomes and costs, to 18 months corrected age, of Family Integrated Care (FICare) for moderate and late preterm infants admitted to a Level II neonatal intensive care unit (NICU). A cluster randomized controlled trial (cRCT) of FICare is currently in progress. FICare is a psycho-educational intervention that empowers parents (mothers and fathers) to sequentially build their knowledge, skill, and confidence so the family is well-prepared to care for their preterm infant before discharge. The FICare cRCT evaluates outcomes related to infant global development and maternal psychosocial distress at 2 months. At 2 months, it is difficult to predict longer term outcomes for moderate and late preterm infants. A follow-up study at 18 months will provide evidence of the sustainability of any effects, and longer-term cost savings upon which to inform policy decisions about full-scale implementation of FICare in Level II NICUs.

DETAILED DESCRIPTION:
Each year, about 15 million of the world's infants are born preterm (<37 weeks gestation), and this number is increasing. In Alberta, the preterm birth rate was 8.43% in 2015, representing 4,749 infants. Alberta has the highest rate of preterm birth among the Canadian provinces, which can be attributed, in part, to delayed child bearing and assisted reproduction. Approximately 20% of all preterm infants are born at <32 weeks GA and require care in a Level III NICU. The remaining 80% are moderate and late preterm infants, which comprises 6.6% of all live births. As gestational age (GA) decreases, the risk of chronic health problems and developmental delays increases. Compared to their full term counterparts, moderate and late preterm infants (born at 32 weeks and zero days [32 0/7] to 36 weeks and six days [36 6/7] GA) are at higher risk for poor health (e.g., increased hospitalizations, respiratory morbidities, and growth and feeding problems) and developmental outcomes (e.g., neurodevelopmental disabilities and cognitive delays, communication and language impairments, and school-related problems). Results of recent studies also indicate that moderate and late preterm infants are at greater risk of experiencing social-emotional problems. In Alberta, preterm infants represent the largest proportion of expenditures of all pediatric health care utilization at 8.45%, with a cost of approximately $35 million per year. The costs associated with preterm infants are greater than for term infants because of longer hospital stays following birth, increased resource utilization, hospital readmissions, and the need for additional health, education, and social services. Financial consequences for families of preterm infants are associated with reduced work force participation and lost earnings, specialized nutritional requirements, and learning and development supports for the child. In addition, there are unquantifiable costs associated with psychological distress, marital and family distress, and social isolation.

The aim of this novel health services research proposal is to assess the longer-term outcomes and costs, to 18 months corrected age, of Family Integrated Care (FICare) for moderate and late preterm infants admitted to a Level II neonatal intensive care unit (NICU). FICare is a psycho-educational intervention that empowers parents (mothers and fathers) to sequentially build their knowledge, skill, and confidence so the family is well-prepared to care for their preterm infant before discharge. FICare is dynamic, whereby parents and healthcare providers openly and mutually negotiate equitable caregiving roles during the infant's NICU stay. Parents are educated and coached to provide routine non-medical care. Healthcare providers continue to provide medical and technical care, such as intravenous medications and procedures, legal documentation, and professional support for families. Using a cluster randomized controlled trial (cRCT) (clinicaltrials.gov ID: NCT02879799), the investigators are evaluating FICare in all 10 Level II NICUs in Alberta (5 intervention, 5 control sites; stratified by hospital size) with follow-up of infant development and costs at age 2 months corrected age. Unless otherwise indicated, infant ages are corrected for prematurity. For the cRCT, investigators hypothesized that FICare would reduce length of NICU stay by 10%, reduce infant morbidities (e.g., nosocomial infections, respiratory support, feeding problems), increase breastmilk feeding, reduce maternal psychological distress, and reduce costs to the health care system and families. Maternal and infant data are currently being collected (1) shortly after admission to the NICU (baseline), (2) shortly before discharge from NICU (outcome), and (3) at 2 months (follow-up). With current funding, investigators can evaluate outcomes related to infant global development and maternal psychosocial distress at 2 months. At 2 months, it is difficult to predict longer term outcomes for moderate and late preterm infants. A follow-up study at 18 months will provide evidence of the sustainability of any effects, and longer-term cost savings upon which to inform policy decisions about full-scale implementation of FICare in Level II NICUs.

The investigators hypothesize that compared to standard care in a Level II NICU, FICare will: (1) improve global development of moderate and late preterm infants at 18 months (primary outcome); (2) improve infant social and emotional development; (3) reduce the frequency of child emergency department visits, hospital readmission rates, and physician visits additional to recommended health surveillance visits; (4) improve child growth trajectories; (5) decrease use of antibiotic prescriptions; (6) increase maternal confidence in caring for their child; (7) decrease maternal psychosocial distress; (8) improve maternal-reported toddler sleep, and (9) decrease public healthcare payer costs.

There is currently no standardized timeline for follow-up of infants born prematurely. Evidence suggests that 18 months is ideal for follow-up because there is decreased inter-individual variability in child development, and social-emotional outcomes can be more accurately assessed. After 18 months, environmental factors may exert a stronger influence on infant development, potentially diluting the ability to directly measure the effect of FICare. Eighteen months is the age at which Canadian Neonatal Follow-Up Network data are collected for infants admitted to a Level III NICU, which will enable comparisons of some outcomes with infants in the Level II NICU FICare Alberta cRCT. There are no plans for further follow-up past 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of infants born between 32 weeks and zero days and 34 weeks and 6 days gestation who enrolled in the FICare Alberta Level II NICU cluster controlled trial (cRCT). The FICare cRCT enrolled mothers of any age who have decision making capacity; mothers who are able to speak, read and understand English well enough to provide informed consent, and complete surveys online or via telephone.

Exclusion Criteria:

* The FICare Alberta Level II NICU cRCT excluded mothers whose infants have serious congenital or chromosomal anomalies that require surgery, or are receiving palliative care; mothers who are not able to communicate in English; mothers with complex social issues.

Min Age: 18 Months | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Global development | At 18-months corrected age
  Ages and Stages Questionnaire, 3rd edition

SECONDARY OUTCOMES:
Infant social and emotional development | At 18-months corrected age
  Ages and Stages Questionnaire:Social-Emotional, 2nd edition; Brief Infant Toddler Social Emotional Assessment
Number of emergency room visits | At 18-months corrected age
  Provincial healthcare administrative databases
Number of re-admissions to hospital | At 18-months corrected age
  Provincial healthcare administrative databases
Number of unplanned visits to physician or other provider | At 18-months corrected age
  Provincial healthcare administrative databases
Number of antibiotic prescriptions | At 18-months corrected age
  Number of antibiotic prescriptions will be compromised of maternal self-report data, and from the infant chart as collected the provincial healthcare provider in Alberta, Canada. A data disclosure agreement has been executed such that AHS Analysts with the Analytics, Data Integration, Measurement & Reporting (DIMR) team will link FICare data with antibiotic prescriptions from infant discharge home to 18 months corrected age. The number antibiotics prescribed will be summed to provide a total number of antibiotic prescriptions.
General self-efficacy in parenting | At 18-months corrected age
  General Self-Efficacy Scale (GSE): A self-administered scale that assesses a general sense of perceived self-efficacy. Self-efficacy as it relates to parenting is addressed by including items in the participant questionnaire related to parenting.
  Responses are made on a 4-point scale. Sum up the responses to all 10 items to yield the final composite score with a range from 10 to 40. There are no sub-scales and no recoding is required. There is no cut-off score, therefore individuals are not categorized as high or low self-efficacious. The GSE score can be correlated with other traits such as anxiety, and depression.
Parenting stress | At 18-months corrected age
  A 36-item scale, captures general parenting stress and three subscales of Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child.
  Responses 1, 2, 3, 7, 8, 9 and 11 are summed for Defensive Responding. Subscale scores are calculated by summing response items 1-12 for Parental Distress, items 13 - 24 for Parent-Child Dysfunctional Interaction, and items 25 - 36 for Difficult Child. Total Stress score is calculated by summing the raw scores of the subscales.
  Raw scores are converted to T scores and percentiles. Normal range for scores is within the 16th to 84th percentiles. Scores in the 85th to 89th percentile are considered high, and scores in the 90th percentile or higher are considered clinically significant.
Maternal-reported toddler sleep | At 18-months corrected age
  Extended Brief Infant Sleep Questionnaire
Direct industry costs (hospital costs, excluding housekeeping, maintenance, planning and physician times). | At 18-months corrected age
  Provincial healthcare administrative databases
State Anxiety | At 18-months corrected age
  Two sub-scales: 1) long-standing quality of trait anxiety (20 items), and 2) the temporary condition of state anxiety (20 items). Items are rated on a 4-point scale. Item scores are added to obtain subtest total scores. Scoring is reversed for anxiety-absent items (19/40 items). Range of scores for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the state anxiety scale. Normative values are available in the manual. Trait anxiety was collected previously in the FICare cRCT (NCT02879799) therefore, only state anxiety will be collected at 18 months.
Depression | At 18-months corrected age
  Centre for Epidemiologic Studies Depression Scale Revised (CESD-R): This scale is a 20 item self-report measure of depression. A 5-point Likert scale measures symptoms of depression in nine different groups as defined by the American Psychiatric Association Diagnostic and Statistical Manual, fifth edition: (1) Sadness; (2) Loss of Interest; (3) Appetite; (4) Sleep; (5) Thinking/Concentration; (6) Guilt; (7) Tired; (8) Movement; and (9) Suicidal Ideation. The total score is calculated as a sum of responses to all 20 questions. The range of possible scores is between 0 and 60.
  Internal consistency (0.92) was high, and the CESD-R is highly correlated with the score for the original CESD (Pearson correlation coefficient 0.89), the latter of which has an internal consistency of 0.85 - 0.90, and test-retest reliability of 0.45 - 0.70.

CONTACTS AND LOCATIONS:
Overall Officials: Abhay Lodha, MD, Principal Investigator — University of Calgary; Khalid Aziz, MD, Principal Investigator — University of Alberta; Vibhuti Shah, MD, Principal Investigator — University of Toronto
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Discussions are underway to draft a data deposition agreement with Secondary Analyses to Generate Evidence (SAGE).

REFERENCES:
- [Background] O'Brien K, Bracht M, Macdonell K, McBride T, Robson K, O'Leary L, Christie K, Galarza M, Dicky T, Levin A, Lee SK. A pilot cohort analytic study of Family Integrated Care in a Canadian neonatal intensive care unit. BMC Pregnancy Childbirth. 2013;13 Suppl 1(Suppl 1):S12. doi: 10.1186/1471-2393-13-S1-S12. Epub 2013 Jan 31. PMID 23445639
- [Background] Benzies KM. Relational Communications Strategies to Support Family-Centered Neonatal Intensive Care. J Perinat Neonatal Nurs. 2016 Jul-Sep;30(3):233-6. doi: 10.1097/JPN.0000000000000195. PMID 27465456
- [Background] Brown J, Ritchie JA. Nurses' perceptions of parent and nurse roles in caring for hospitalized children. Child Health Care. 1990 Winter;19(1):28-36. doi: 10.1207/s15326888chc1901_4. PMID 10106396
- [Background] Mento G, Nosarti C. The case of late preterm birth: sliding forwards the critical window for cognitive outcome risk. Transl Pediatr. 2015 Jul;4(3):214-8. doi: 10.3978/j.issn.2224-4336.2015.06.02. PMID 26835378
- [Background] Hack M, Wilson-Costello D. Follow-up outcomes of high risk infants. In: Buonocore G, Bracci R, Weindling M, eds. Neonatology: A practical approach to neonatal diseases: Springer; 2012:122-129.
- [Background] March of Dimes, PMNCH, Save the Children, WHO. Born too soon: The global action report on preterm birth. Geneva: World Health Organization;2012.
- [Background] World Health Organization. Preterm birth fact sheet. 2015; www.who.int/mediacentre/factsheets/fs363/en.
- [Background] Alberta Health and Wellness. Interactive Health Data Application, 2015 reproductive health data set. 2015; www.ahw.gov.ab.ca/IHDA_Retrieval/selectSubCategoryParameters.do#.
- [Background] Canadian Institute for Health Information. Highlights of 2010-2011 selected indicators describing the birthing process in Canada. Canadian Institute for Health Information;2012.
- [Background] Tough SC, Newburn-Cook C, Johnston DW, Svenson LW, Rose S, Belik J. Delayed childbearing and its impact on population rate changes in lower birth weight, multiple birth, and preterm delivery. Pediatrics. 2002 Mar;109(3):399-403. doi: 10.1542/peds.109.3.399. PMID 11875131
- [Background] Tough S, Tofflemire K, Newburn-Cook C, Fraser-Lee N, Benzies K. Increased risks of pregnancy complications and adverse infant outcomes associated with assisted reproduction. International Congress Series. Research Papers in Fertility and Reproductive Medicine. Proceedings of the 18th World Congress on Fertility and Sterility (IFFS 2004). 2004;1271:376-379.
- [Background] Kerstjens JM, de Winter AF, Bocca-Tjeertes IF, Bos AF, Reijneveld SA. Risk of developmental delay increases exponentially as gestational age of preterm infants decreases: a cohort study at age 4 years. Dev Med Child Neurol. 2012 Dec;54(12):1096-101. doi: 10.1111/j.1469-8749.2012.04423.x. Epub 2012 Sep 30. PMID 23020259
- [Background] Tomashek KM, Shapiro-Mendoza CK, Davidoff MJ, Petrini JR. Differences in mortality between late-preterm and term singleton infants in the United States, 1995-2002. J Pediatr. 2007 Nov;151(5):450-6, 456.e1. doi: 10.1016/j.jpeds.2007.05.002. Epub 2007 Jul 24. PMID 17961684
- [Background] Sun Y, Hsu P, Vestergaard M, Christensen J, Li J, Olsen J. Gestational age, birth weight, and risk for injuries in childhood. Epidemiology. 2010 Sep;21(5):650-7. doi: 10.1097/EDE.0b013e3181e94253. PMID 20585254
- [Background] Schonhaut L, Armijo I, Perez M. Gestational age and developmental risk in moderately and late preterm and early term infants. Pediatrics. 2015 Apr;135(4):e835-41. doi: 10.1542/peds.2014-1957. Epub 2015 Mar 2. PMID 25733752
- [Background] Engle WA; American Academy of Pediatrics Committee on Fetus and Newborn. Age terminology during the perinatal period. Pediatrics. 2004 Nov;114(5):1362-4. doi: 10.1542/peds.2004-1915. PMID 15520122
- [Background] Harijan P, Boyle EM. Health outcomes in infancy and childhood of moderate and late preterm infants. Semin Fetal Neonatal Med. 2012 Jun;17(3):159-62. doi: 10.1016/j.siny.2012.02.002. Epub 2012 Mar 13. PMID 22417643
- [Background] Baron IS, Litman FR, Ahronovich MD, Baker R. Late preterm birth: a review of medical and neuropsychological childhood outcomes. Neuropsychol Rev. 2012 Dec;22(4):438-50. doi: 10.1007/s11065-012-9210-5. Epub 2012 Aug 7. PMID 22869055
- [Background] McGowan JE, Alderdice FA, Holmes VA, Johnston L. Early childhood development of late-preterm infants: a systematic review. Pediatrics. 2011 Jun;127(6):1111-24. doi: 10.1542/peds.2010-2257. Epub 2011 May 29. PMID 21624885
- [Background] Johnson S, Evans TA, Draper ES, Field DJ, Manktelow BN, Marlow N, Matthews R, Petrou S, Seaton SE, Smith LK, Boyle EM. Neurodevelopmental outcomes following late and moderate prematurity: a population-based cohort study. Arch Dis Child Fetal Neonatal Ed. 2015 Jul;100(4):F301-8. doi: 10.1136/archdischild-2014-307684. Epub 2015 Apr 1. PMID 25834170
- [Background] Guy A, Seaton SE, Boyle EM, Draper ES, Field DJ, Manktelow BN, Marlow N, Smith LK, Johnson S. Infants born late/moderately preterm are at increased risk for a positive autism screen at 2 years of age. J Pediatr. 2015 Feb;166(2):269-75.e3. doi: 10.1016/j.jpeds.2014.10.053. Epub 2014 Dec 2. PMID 25477165
- [Background] Kerstjens JM, de Winter AF, Bocca-Tjeertes IF, ten Vergert EM, Reijneveld SA, Bos AF. Developmental delay in moderately preterm-born children at school entry. J Pediatr. 2011 Jul;159(1):92-8. doi: 10.1016/j.jpeds.2010.12.041. Epub 2011 Feb 16. PMID 21324481
- [Background] Ballantyne M, Benzies KM, McDonald S, Magill-Evans J, Tough S. Risk of developmental delay: Comparison of late preterm and full term Canadian infants at age 12 months. Early Hum Dev. 2016 Oct;101:27-32. doi: 10.1016/j.earlhumdev.2016.04.004. Epub 2016 Jul 9. PMID 27405053
- [Background] Stene-Larsen K, Brandlistuen RE, Lang AM, Landolt MA, Latal B, Vollrath ME. Communication impairments in early term and late preterm children: a prospective cohort study following children to age 36 months. J Pediatr. 2014 Dec;165(6):1123-8. doi: 10.1016/j.jpeds.2014.08.027. Epub 2014 Sep 23. PMID 25258153
- [Background] Chan E, Quigley MA. School performance at age 7 years in late preterm and early term birth: a cohort study. Arch Dis Child Fetal Neonatal Ed. 2014 Nov;99(6):F451-7. doi: 10.1136/archdischild-2014-306124. Epub 2014 Jun 25. PMID 24966128
- [Background] de Jong M, Verhoeven M, van Baar AL. School outcome, cognitive functioning, and behaviour problems in moderate and late preterm children and adults: a review. Semin Fetal Neonatal Med. 2012 Jun;17(3):163-9. doi: 10.1016/j.siny.2012.02.003. Epub 2012 Feb 23. PMID 22364677
- [Background] van Baar AL, Vermaas J, Knots E, de Kleine MJ, Soons P. Functioning at school age of moderately preterm children born at 32 to 36 weeks' gestational age. Pediatrics. 2009 Jul;124(1):251-7. doi: 10.1542/peds.2008-2315. PMID 19564307
- [Background] Hornman J, de Winter AF, Kerstjens JM, Bos AF, Reijneveld SA. Emotional and Behavioral Problems of Preterm and Full-Term Children at School Entry. Pediatrics. 2016 May;137(5):e20152255. doi: 10.1542/peds.2015-2255. PMID 27244786
- [Background] Potijk MR, de Winter AF, Bos AF, Kerstjens JM, Reijneveld SA. Higher rates of behavioural and emotional problems at preschool age in children born moderately preterm. Arch Dis Child. 2012 Feb;97(2):112-7. doi: 10.1136/adc.2011.300131. Epub 2011 Dec 6. PMID 22147746
- [Background] Potijk MR, de Winter AF, Bos AF, Kerstjens JM, Reijneveld SA. Co-occurrence of developmental and behavioural problems in moderate to late preterm-born children. Arch Dis Child. 2016 Mar;101(3):217-22. doi: 10.1136/archdischild-2015-308958. Epub 2015 Oct 15. PMID 26471109
- [Background] Blaggan S, Guy A, Boyle EM, Spata E, Manktelow BN, Wolke D, Johnson S. A parent questionnaire for developmental screening in infants born late and moderately preterm. Pediatrics. 2014 Jul;134(1):e55-62. doi: 10.1542/peds.2014-0266. PMID 24982100
- [Background] Johnson S, Matthews R, Draper ES, Field DJ, Manktelow BN, Marlow N, Smith LK, Boyle EM. Early Emergence of Delayed Social Competence in Infants Born Late and Moderately Preterm. J Dev Behav Pediatr. 2015 Nov-Dec;36(9):690-9. doi: 10.1097/DBP.0000000000000222. PMID 26461097
- [Background] Dean S. Child Health Strategic Clinical Network meeting: Reporting and analytics. Calgary, AB: Alberta Health Services; 2012.
- [Background] Petrou S, Khan K. Economic costs associated with moderate and late preterm birth: primary and secondary evidence. Semin Fetal Neonatal Med. 2012 Jun;17(3):170-8. doi: 10.1016/j.siny.2012.02.001. Epub 2012 Feb 23. PMID 22364679
- [Background] Briggs-Gowan MJ, Carter AS, Irwin JR, Wachtel K, Cicchetti DV. The Brief Infant-Toddler Social and Emotional Assessment: screening for social-emotional problems and delays in competence. J Pediatr Psychol. 2004 Mar;29(2):143-55. doi: 10.1093/jpepsy/jsh017. PMID 15096535
- [Background] Kolb B, Whishaw IQ, Teskey GC. An introduction to brain and behavior. New York, NY: Worth Publishers; 2016.
- [Background] Shulruf B, Morton S, Goodyear-Smith F, O'Loughlin C, Dixon R. Designing multidisciplinary longitudinal studies of human development: analyzing past research to inform methodology. Eval Health Prof. 2007 Sep;30(3):207-28. doi: 10.1177/0163278707304030. PMID 17693616
- [Background] Scher MS, Johnson MW, Ludington SM, Loparo K. Physiologic brain dysmaturity in late preterm infants. Pediatr Res. 2011 Nov;70(5):524-8. doi: 10.1203/PDR.0b013e31822f24af. PMID 21796018
- [Background] Schwichtenberg AJ, Christ S, Abel E, Poehlmann-Tynan JA. Circadian Sleep Patterns in Toddlers Born Preterm: Longitudinal Associations with Developmental and Health Concerns. J Dev Behav Pediatr. 2016 Jun;37(5):358-69. doi: 10.1097/DBP.0000000000000287. PMID 27011003
- [Background] Booker CL, Harding S, Benzeval M. A systematic review of the effect of retention methods in population-based cohort studies. BMC Public Health. 2011 Apr 19;11:249. doi: 10.1186/1471-2458-11-249. PMID 21504610
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy Scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Casual and control beliefs (pp. 35-37). Windsor, UK: NFER-NELSON.
- [Background] Eaton WW, Muntaner C, Smith C, Tien A, Ybarra M. Center for Epidemiologic Studies Depression Scale: Review and revision (CESD and CESD-R). In: Maruish ME, ed. The Use of Psychological Testing for Treatment Planning and Outcomes Assessment. 3rd ed. Mahwah, NJ: Lawrence Erlbaum; 2004:363-377.
- [Background] Sadeh A, Mindell JA, Luedtke K, Wiegand B. Sleep and sleep ecology in the first 3 years: a web-based study. J Sleep Res. 2009 Mar;18(1):60-73. doi: 10.1111/j.1365-2869.2008.00699.x. Epub 2008 Oct 16. PMID 19021850
- [Background] Sadeh A. A brief screening questionnaire for infant sleep problems: validation and findings for an Internet sample. Pediatrics. 2004 Jun;113(6):e570-7. doi: 10.1542/peds.113.6.e570. PMID 15173539
- [Background] Sadeh A, Mindell J, Rivera L. "My child has a sleep problem": a cross-cultural comparison of parental definitions. Sleep Med. 2011 May;12(5):478-82. doi: 10.1016/j.sleep.2010.10.008. Epub 2011 Apr 7. PMID 21478050
- [Background] Radloff, L. S. (1977). The CES-D scale: A self report depression scale for research in the general population. Applied Psychological Measurements, 1, 385-401.
- [Background] Teng A, Bartle A, Sadeh A, Mindell J. Infant and toddler sleep in Australia and New Zealand. J Paediatr Child Health. 2012 Mar;48(3):268-73. doi: 10.1111/j.1440-1754.2011.02251.x. Epub 2011 Nov 22. PMID 22107168
- [Background] Mindell JA, Du Mond CE, Sadeh A, Telofski LS, Kulkarni N, Gunn E. Efficacy of an internet-based intervention for infant and toddler sleep disturbances. Sleep. 2011 Apr 1;34(4):451-8. doi: 10.1093/sleep/34.4.451. PMID 21461323
- [Background] Caro J, Erslev AJ. Uremic inhibitors of erythropoiesis. Semin Nephrol. 1985 Jun;5(2):128-32. No abstract available. PMID 3879951
- [Background] Spielberger CD, Gorsuch RL, Lushene RE. Test manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press; 1970.
- [Background] Abidin RR. Parenting Stress Index - Fourth Edition - Short Form. Lutz, FL: Psychological Assessment Resources; 2012.
- [Background] Eaton WW, Smith C, Ybarra M, Muntaner C, Tien A. Center for Epidemiologic Studies Depression Scale: Review and revision (CESD and CESD-R). In: Maruish ME, ed. The use of psychological testing for treatment planning and outcomes assessment: Volume 3 - Instruments for adults. Mahwah, NJ: Lawrence Erlbaum Associates; 2004:363-377.
- [Background] Schwarzer R, Jerusalem M. Generalized Self-Efficacy Scale. In: Weinman J, Wright S, Johnston M, eds. Measures in health psychology: A user's portfolio. Causal and control beliefs. Windsor, UK: NEFR-NELSON; 1995:35-37.